CLINICAL TRIAL: NCT05080413
Title: Comparison of Sensory Cuing Modalities for Freezing of Gait in Patients With Idiopathic Parkinson's Disease : a Pilot Study
Brief Title: Comparison of Sensory Cuing Modalities for Freezing of Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Health Service Medical Center, Seoul, Korea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-08-025
Record Dates: First submitted 2021-09-14; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait; Parkinson Disease; functional near-infrared spectroscopy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study is a single group pre-post intervention comparison study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson disease group (Experimental): A total of 10 patients in this group will walk under the same conditions (off- state of antiparkinson drugs). Participants will be instructed to walk three laps on a 10-meter track under each of the following three conditions : 1) without stimulation, 2) with visual cues using a laser shoe, 3) with auditory cues using a metronome.
  Interventions: Device: Laser shoes; Device: Metronome

INTERVENTIONS:
Device: Laser shoes — Path Finder® is a device that is fixed to the noses of the patient's shoes using a rubber strap, and laser-marks the place to be stepped on the ground of the opposite foot when walking. It is installed on both feet to relieve the symptoms of freezing of gait.
  Other Names: Path Finder®
Device: Metronome — The metronome, which makes a sound with a constant beat, is known to have an effect on the symptoms of Freezing of Gait in Parkinson's disease patients. At a rate of 80 beats per minute, the volume of sound that the patient can fully recognize is set to resolve the freezing of gait using the metronome sound.

SUMMARY:
The investigators intend to compare the effects on the resolution of visual and auditory sensory cues on the resolution of freezing of gait in patients with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
As Parkinson's disease progresses, the patients develop 'Freezing of gait', which make it difficult to initiate gait, turn at the corner, and enter a narrow space. This is considered to be a very important symptom, as it is related to the performance of daily activities, independence of life, and serious injuries caused by falls while walking in Parkinson's disease patients.

It has been found that the use of external sensory stimulation (visual, auditory) can reduce the symptoms of Freezing of Gait, and is used as rehabilitation treatment and instant symptomatic resolution. However, the relative effectiveness of sensory stimulation is not studied yet.

Accordingly, the investigators intend to compare the effects of visual and auditory sensory cues on the resolution of freezing of gait in patients with idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic Parkinson's disease with freezing of gait according to the United Kingdom (UK) Brain Bank.
2. Scored more than 15 points of Korean version of mini-mental status exam (K-MMSE).
3. Independent gait for at least a minute without walking assistance device.

Exclusion Criteria:

1. History of concomitant brain disease other than idiopathic Parkinson's disease.
2. Other neurologically deteriorated states, such as neuromuscular disease, which can cause gait disturbance.
3. Other psychiatric disorders.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-28 (Actual)

PRIMARY OUTCOMES:
Number of freezing of gait episodes | 30 minutes
  The number of occurrences of freezing of gait will be measured in each of the three situations (no sensory stimulation, visual stimulation, and auditory stimulation).
Duration of freezing of gait episodes | 30 minutes
  The average duration per occurrence of freezing of gait in each of the three situations (no sensory stimulation, visual stimulation, and auditory stimulation) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yup Kim, M.D., Principal Investigator — Veterans Health Service Medical Center, Seoul, Korea
Locations (1):
- Veterans Health Service Medical Center, Seoul, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers.

REFERENCES:
- [Background] Bartels AL, Leenders KL. Parkinson's disease: the syndrome, the pathogenesis and pathophysiology. Cortex. 2009 Sep;45(8):915-21. doi: 10.1016/j.cortex.2008.11.010. Epub 2008 Nov 27. PMID 19095226
- [Background] Heremans E, Nieuwboer A, Vercruysse S. Freezing of gait in Parkinson's disease: where are we now? Curr Neurol Neurosci Rep. 2013 Jun;13(6):350. doi: 10.1007/s11910-013-0350-7. PMID 23625316
- [Background] Shine JM, Naismith SL, Lewis SJ. The pathophysiological mechanisms underlying freezing of gait in Parkinson's Disease. J Clin Neurosci. 2011 Sep;18(9):1154-7. doi: 10.1016/j.jocn.2011.02.007. Epub 2011 Jul 2. PMID 21724402
- [Background] Gao C, Liu J, Tan Y, Chen S. Freezing of gait in Parkinson's disease: pathophysiology, risk factors and treatments. Transl Neurodegener. 2020 Apr 15;9:12. doi: 10.1186/s40035-020-00191-5. eCollection 2020. PMID 32322387
- [Background] Lee SJ, Yoo JY, Ryu JS, Park HK, Chung SJ. The effects of visual and auditory cues on freezing of gait in patients with Parkinson disease. Am J Phys Med Rehabil. 2012 Jan;91(1):2-11. doi: 10.1097/PHM.0b013e31823c7507. PMID 22157432
- [Background] Barthel C, Nonnekes J, van Helvert M, Haan R, Janssen A, Delval A, Weerdesteyn V, Debu B, van Wezel R, Bloem BR, Ferraye MU. The laser shoes: A new ambulatory device to alleviate freezing of gait in Parkinson disease. Neurology. 2018 Jan 9;90(2):e164-e171. doi: 10.1212/WNL.0000000000004795. Epub 2017 Dec 20. PMID 29263221
- [Background] Arias P, Cudeiro J. Effect of rhythmic auditory stimulation on gait in Parkinsonian patients with and without freezing of gait. PLoS One. 2010 Mar 22;5(3):e9675. doi: 10.1371/journal.pone.0009675. PMID 20339591
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Derived] An EJ, Sim WS, Kim SM, Kim JY. Suitability of visual cues for freezing of gait in patients with idiopathic Parkinson's disease: a case-control pilot study. J Neuroeng Rehabil. 2023 Jul 18;20(1):91. doi: 10.1186/s12984-023-01214-8. PMID 37464390